CLINICAL TRIAL: NCT05544149
Title: An Open-label, Phase II Single Arm Trial of Thoracic Radiotherapy for?ES-SCLC After First Line Treatment With Immune Checkpoint Inhibitors
Brief Title: TRT for ES-SCLC After First Line Treatment With Immune Checkpoint Inhibitors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiaojing Lai, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-TRT-SCLC-IIT
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: SCLC,Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRT (Experimental): Patients with es-SCLC after first line treatment with immune checkpoint inhibitors will be treated with thoracic radiotherapy.
  Interventions: Radiation: Thoracic radiotherapy

INTERVENTIONS:
Radiation: Thoracic radiotherapy — Thoracic radiotherapy for ES-SCLC after first line immunecheckpoint inhibitors

SUMMARY:
To Evaluate the Safety and Efficacy of Thoracic Radiotherapy for?ES-SCLC After First Line Treatment with Immune Checkpoint Inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* ECOG PS 0-1.
* Histological or cytological syndrome of small cell lung cancer, imaging evaluation staging is extensive
* Life expectancy >= 3 months.
* Patients are non-progressed after 4 dosed of immunotherapy plus platinum based chemotherapy, with residual thoracic lesions
* Palliative radiotherapy were allowed except for TRT, the interval > 4 weeks
* Adequate organ function prior to enrollment:
* Adequate bone marrow function: white blood cell (WBC) count ≥ 3.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, platelet count ≥ 100 * 10 ^ 9/L and hemoglobin ≥90g/L,;
* Adequate hepatic function: total bilirubin, urea nitrogen and serum creatinine≤ 1.5 x upper limit of normal (ULN). Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.0 ULN;
* Sufficient heart and lung function, EF>55%FEV1>50%
* Ability to understand and willingness to provide the informed consent.
* Women of childbearing age and men must agree to use effective contraception during the trial.

Exclusion Criteria:

* History of another malignancy or concurrent malignancy;
* Mixed small cell with non-small cell lung cancer histology;
* History of thoracic radiotherapy;
* Malignant pleural or ascites;
* Patients with leptomeningeal metastasis or uncontrolled brain;
* Severe autoimmune disease: inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Wegener's granulomatosis and related vasculitides.
* Symptomatic interstitial lung disease or clinically active infectious/non-infectious pneumonitis.
* Active infection, congestive heart failure, or any evidence of myocardial infarction, unstable angina pectoris or cardiac arrhythmia within 6 months prior to enrollment.
* The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival | 2 years
  From the date of enrollment to the date of local recurrence
Adverse events | 2 years
  Treatment-related adverse events according to CTCAE 5.0.

SECONDARY OUTCOMES:
Progress free survival | 2 years
  From the date of enrollment to the date of disease progression
Overall survival | 2 years
  from the date of enrollment until death by any cause or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Lai, Principal Investigator — Department of Thoracic Radiotherapy, Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No